CLINICAL TRIAL: NCT02931136
Title: Early Diagnosis and Early Treatment of Alzheimer's Disease Based on Senile Plaque Imaging
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, xiaoshifu, Director, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Shanghai Mental Health Center
Record Dates: First submitted 2016-10-08; First posted 2016-10-12 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Mild Cognitive Impairment; Biomarker; Diagnosis; Treatment
MeSH Terms: conditions — Cognitive Dysfunction; Disease | interventions — huperzine A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): Huperzine A treatment.
  Interventions: Drug: Huperzine A
- Placebo group (Placebo Comparator): The placebo in 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Huperzine A — The participants will treatment by the Huperzine A 200 ug/day in 52 weeks.
  Other Names: shuang yi ping
  Arms: treatment group
Drug: Placebo — The participants will treatment by the placebo in 52 weeks.
  Arms: Placebo group

SUMMARY:
The purpose of this study is based on the Flutemetamol-PET senile plaque imaging to investigate the peripheral blood biochemical and brain MRI imaging biomarkers and to research completely independent intellectual property rights neuropsychological test tool for the MCI due to AD. At the same time, the investigators will study the efficacy and safety of early treatment of MCI due to AD by Huperzine A in 52 weeks.

DETAILED DESCRIPTION:
This is a randmized, double-blind, placebo-controll study.

ELIGIBILITY:
Inclusion Criteria:

* memory complaint, preferably corroborated by a spouse or relative.
* objective memory impairment.
* normal general cognitive function.
* intact activities of daily living.
* absence of dementia.
* the positive of brain senile plaque.

Exclusion Criteria:

* more than two lacuna ischemia (of diameter < 1 cm) as revealed by MRI fluid-attenuated inversion recovery (FLAIR) sequence.
* other type of dementia except AD

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The average annual conversion rate in patients of MCI due to AD convert to the AD. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shifu Xiao, M.D., Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes